CLINICAL TRIAL: NCT07129200
Title: The Effects of Caffeine Supplementation on Exercise Physiology and Time-trial Performance in a Hot Environment
Brief Title: The Effects of Caffeine on Exercise Physiology and Time-trial Performance in a Hot Environment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Mary's University, Twickenham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: SMU_ETHICS_2024-25_1111
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Caffeine; Thermoregulation
Keywords: caffeine; thermoregulation; time trial; exercise physiology

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caffeine (Experimental): 5 mg/kg dose of caffeine (in pill form)
  Interventions: Other: Hot environment; Other: Thermoneutral environment
- Placebo (Placebo Comparator): 5 mg/kg dose of placebo (maltodextrin - in pill form)
  Interventions: Other: Hot environment; Other: Thermoneutral environment

INTERVENTIONS:
Other: Hot environment — Hot environment of 35 degrees Celsius
Other: Thermoneutral environment — Thermoneutral environment of 18 degrees Celsius

SUMMARY:
Maintaining a stable core temperature is vital for physiological function; yet, exercise in heat can be problematic, and there is risk of exertional heat-related illness (Flouris & Schlader, 2015; Leyk et al., 2019; Périard et al., 2021; Tyler et al., 2016; Veltmeijer et al., 2015). While aerobic fitness improves heat tolerance (Alhadad et al., 2019), strategies like acclimation and pre-cooling also mitigate heat stress (Casadio et al., 2016; Lorenzo et al., 2010; Ross et al., 2013; Siegel et al., 2010). Caffeine, an ergogenic aid (Del Corso et al., 2011; John et al., 2024), is known to enhance performance via adenosine antagonism and increased catecholamines in normothermic environments (Fredholm et al., 1999; Graham & Spriet, 1991). However, effects in heat are inconsistent (Ganio et al., 2009; Zhang et al., 2014), possibly due to caffeine reducing the ability to thermoregulate effectively. Therefore, the aim of this study is to investigate the effects of a moderate dose of caffeine (5 mg/kg) on thermoregulation during a 30-minute running time trial in 35°C heat.

ELIGIBILITY:
Inclusion Criteria:

* Healthy trained runners

Exclusion Criteria:

-

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-08-22 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Blood lactate concentration | From baseline to completion, up to 31 days
  Change from baseline in blood lactate concentration measured at rest and at five different exercise intensities (65, 70, 75, 80, and 85% percent of maximal oxygen uptake) on a treadmill.
Heart rate | From baseline to completion, up to 31 days
  Change from baseline in heart rate measured at rest and at five different exercise intensities (65, 70, 75, 80, and 85% percent of maximal oxygen uptake) on a treadmill.
Rating of perceived exertion | From baseline to completion, up to 31 days
  Change from baseline in rating of perceived exertion measured (using the 6-20 Borg scale) at five different exercise intensities (65, 70, 75, 80, and 85% percent of maximal oxygen uptake) on a treadmill.
Oxygen uptake | From baseline to completion, up to 31 days
  Change from baseline in oxygen uptake measured at five different exercise intensities (65, 70, 75, 80, and 85% percent of maximal oxygen uptake) on a treadmill.
Time trial performance | From baseline to completion, up to 31 days
  Change from baseline in distance covered during a 30 minute time trial on a treadmill.